CLINICAL TRIAL: NCT00436410
Title: An Evaluation of the Tissue Distribution and the Selective Tumor Trafficking of TNF-Bound Colloidal Gold (CYT-6091) Following Intravenous Administration in Subjects With Primary and Metastatic Cancer Undergoing Surgical Resection
Brief Title: Tumor Necrosis Factor in Patients Undergoing Surgery for Primary Cancer or Metastatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 070043; 07-C-0043; NCI-P6066; CYT-NCI-07-C-0043; CDR0000529849
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Adrenocortical Carcinoma; Breast Cancer; Colorectal Cancer; Gastrointestinal Cancer; Kidney Cancer; Liver Cancer; Melanoma (Skin); Ovarian Cancer; Pancreatic Cancer; Sarcoma
Keywords: stage IV colon cancer; stage IV rectal cancer; adult primary hepatocellular carcinoma; stage IV pancreatic cancer; male breast cancer; stage IV breast cancer; stage IV melanoma; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer; recurrent adrenocortical carcinoma; stage I adrenocortical carcinoma; stage II adrenocortical carcinoma; stage III adrenocortical carcinoma; stage IV adrenocortical carcinoma; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; advanced adult primary liver cancer; localized resectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent melanoma; stage I melanoma; stage II melanoma; stage III melanoma; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; recurrent ovarian epithelial cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; gastrointestinal cancer; adult fibrosarcoma; recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Adrenocortical Carcinoma; Breast Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Kidney Neoplasms; Liver Neoplasms; Melanoma; Ovarian Neoplasms; Pancreatic Neoplasms; Sarcoma; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular; Breast Neoplasms, Male; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Fibrosarcoma | interventions — CYT-6091; Microscopy, Electron

INTERVENTIONS:
Biological: colloidal gold-bound tumor necrosis factor
Other: electron microscopy
Other: pharmacological study
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies, such as tumor necrosis factor, may stimulate the immune system in different ways and stop tumor cells from growing. Studying tumor necrosis factor in samples of tumor tissue and healthy tissue from patients with cancer in the laboratory may help doctors learn how tumor necrosis factor works in tumor tissue and healthy tissue.

PURPOSE: This clinical trial is studying tumor necrosis factor in patients undergoing surgery for primary cancer or metastatic cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the tumor tissue and normal tissue distribution of colloidal gold-bound tumor necrosis factor in patients with primary or metastatic cancer undergoing surgery.

Secondary

* Determine, by histological examination of resected tumor tissue, the acute antitumor effects of this treatment in these patients.
* Determine the long-term toxicities of this treatment in these patients.
* Determine the response to this treatment in these patients.

OUTLINE: This is a cohort study. Patients are stratified according to disease type (colorectal cancer vs hepatocellular cancer vs pancreatic exocrine cancer vs pancreatic endocrine cancer vs breast cancer vs melanoma vs primary adrenal tumors vs renal cell carcinoma).

Patients receive colloidal gold-bound tumor necrosis factor IV over 15-30 seconds 12-78 hours prior to surgery. Patients then undergo standard-care surgery.

Tumor and normal tissues are removed during surgery for analysis of antitumor effects and tissue distribution of colloidal gold-bound tumor necrosis factor by electron microscopy.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 108 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or metastatic malignancy, including any of the following:

  * Colorectal cancer
  * Hepatocellular cancer
  * Pancreatic exocrine cancer
  * Pancreatic endocrine cancer
  * Breast cancer
  * Melanoma
  * Sarcoma
  * Primary adrenal tumors
  * Renal cell carcinoma
  * Ovarian cancer
  * Adenocarcinoma of gastrointestinal origin
  * Peritoneal mesothelioma
* Clinical indication for surgical resection
* No known brain metastases

  * Previously treated brain metastases with no evidence of recurrence allowed
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 5 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.5 mg/dL
* ALT and AST ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Hemoglobin ≥ 9.0 g/dL
* Ejection fraction ≥ 45% by echocardiogram, thallium stress test, or MUGA (for patients with prior cardiovascular disease)
* FEV_1 OR DLCO > 30% of predicted (for patients with prior pulmonary disease)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active bacterial infection

  * Localized chronic infection (e.g., mild acne, tinea pedis) allowed
* No known bleeding disorder
* No other serious illness including, but not limited to, any of the following:

  * Unstable angina
  * Severe oxygen-dependent chronic obstructive pulmonary disease
  * End-stage liver disease
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy, including cytotoxic drugs, radiotherapy, surgery, or other anticancer modalities
* More than 3 weeks since prior biologic therapy or cytotoxic agents (6 weeks for nitrosoureas) and recovered
* No concurrent treatment in a protocol for which patient is being evaluated for response
* No other concurrent anticancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2006-12; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Tumor tissue and normal tissue distribution of colloidal gold-bound tumor necrosis factor
Comparison of the impact of distribution time and histology on accumulation of treatment particles in tumor vs normal tissues

SECONDARY OUTCOMES:
Acute antitumor activity of treatment
Long-term toxicity of treatment as assessed by CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - NCI - Center for Cancer Research-Medical Oncology, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland

REFERENCES:
- [Derived] Kesharwani P, Ma R, Sang L, Fatima M, Sheikh A, Abourehab MAS, Gupta N, Chen ZS, Zhou Y. Gold nanoparticles and gold nanorods in the landscape of cancer therapy. Mol Cancer. 2023 Jun 21;22(1):98. doi: 10.1186/s12943-023-01798-8. PMID 37344887